CLINICAL TRIAL: NCT05636475
Title: The Effect Of Machine-Based And Manually Applied Hand Massage On Pain, Anxiety And Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Münevver Şengül (Other)
Collaborators: Bartin State Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Münevver Şengül, Sponsor Investigator, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-SBB-0329
Record Dates: First submitted 2022-11-07; First posted 2022-12-05 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Laparoscopic cholecystectomy; hand massage; postoperative anxiety; postoperative pain; gastrointestinal tract function; machine-based
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manuel hand massage group (Experimental): According to the hand massage training received, the patient coming out of the surgery is in diamond shape for ten minutes for each hand.
  Interventions: Other: Manual hand massage after laparoscopic cholecystectomy surgery
- machine-based hand massage (Experimental): The pressure setting of the machine is made according to the manual massage application method. In manual massage and machine massage, machine adjustments are made to keep the temperature and pressure difference as low as possible. A hand massage is done for ten minutes for each hand.
  Interventions: Other: Machine-based hand massage after laparoscopic cholecystectomy surgery
- Control group (No Intervention): The control group will be treated only according to the clinical analgesia protocol.

INTERVENTIONS:
Other: Manual hand massage after laparoscopic cholecystectomy surgery — Manual hand massage is applied to a group of patients at 0, 4 and 8 hours after the patient returns from laparoscopic cholecystectomy surgery. It is applied to each hand for ten minutes.
  Arms: Manuel hand massage group
Other: Machine-based hand massage after laparoscopic cholecystectomy surgery — Machine-based hand massage is applied to a group of patients at 0, 4 and 8 hours after the patient returns from laparoscopic cholecystectomy surgery. It is applied to each hand for ten minutes.
  Arms: machine-based hand massage

SUMMARY:
Introduction: As after almost every surgical procedure, changes in the patient's system functions, acute pain and an increase in anxiety level occur after laparoscopic cholecystectomy. Uncontrolled pain and anxiety slows down the healing process, increases the possibility of opioid use and the risk of undesirable side effects, and increases mortality, and prolongs hospital discharge.

Objective: The aim of the thesis study is to evaluate the effect of machine-based and manual hand massage applied in the postoperative period on pain, anxiety and gastrointestinal system functions in patients who have undergone laparoscopic cholecystectomy.

Method: In the study planned as a randomized controlled experimental study; There will be 3 groups, 57 patients in each group, including the experimental groups and the control group, who have undergone laparoscopic cholecystectomy and hospitalized in the General Surgery Clinic of Bartın State Hospital, where machine-based and manual hand massage will be applied. In addition to the analgesic treatment requested by the physician at the 0th, 4th and 8th hours after the surgery, the experimental groups will be given 10 minutes of hand massage to each hand, and only the requested treatment will be applied to the control group. After the applications, the changes in the pain and anxiety levels of the patients as well as the effects on the gastrointestinal system functions will be recorded. 'Data Collection Form', 'Numerical Rating Scale', 'State-Trait Anxiety Scale' and 'Gastrointestinal functions monitoring form' will be used to collect the data and the data will be analyzed in SPSS 22.0 program.

DETAILED DESCRIPTION:
As with almost every surgical procedure, changes in the patient's system functions, acute pain and an increase in anxiety level occur after laparoscopic cholecystectomy. Uncontrolled pain and anxiety slows down the healing process, increases the possibility of opioid use and the risk of undesirable side effects, and increases mortality, and prolongs hospital discharge. Massage; increases patient comfort, relaxation and satisfaction and reduces stress. Receptors associated with nerve fibers that transmit pain to the brain are mostly found in the feet and hands. For this reason, the effect of hand massage was wanted to be examined.

The aim of the thesis study is to evaluate the effect of manual and machine-based application of hand massage on pain, anxiety and GIS functions after laparoscopic cholecystectomy. In the study planned as a randomized controlled experimental study; There will be 3 groups, 57 patients in each group, including the experimental groups and the control group, who have undergone laparoscopic cholecystectomy and hospitalized in the General Surgery Clinic of Bartın State Hospital, where machine-based and manual hand massage will be applied.

First, the researcher will receive certified training on hand massage. Necessary permissions will be obtained to carry out the research. Patients who have undergone laparoscopic cholecystectomy in the general surgery service of Bartın state hospital and meet the inclusion criteria will be divided into 3 groups, 2 experimental and 1 control group, by block randomization. Before starting the application, the purpose of the research will be explained by the researcher and the informed consent of the individuals will be obtained. Data will be collected between September 2022 and June 2023. The patient will fill in the 'Section 1 of the Data Collection Form' and the 'Trait Anxiety Scale' at least 1 hour before the surgery in the preoperative period. The second part will be filled at the most appropriate time after the surgery. When the patient comes to the service after the surgery, before the first hour is up, that is, at the 0th hour and at the 4th and 8th hours, a hand massage device will be used and manual hand massage will be applied in addition to the treatment according to the clinical analgesia protocol, and hand massage will be applied for 10 minutes for each hand. The control group will be treated only according to the clinical analgesia protocol. Before the massage and after the massage at 0, 4 and 8 hours; On the other hand, the 'Numerical Rating Scale', State Anxiety Scale' will be applied to the control group during the periods when other groups are massaged without hand massage, and the 'Gastrointestinal Functions Monitoring Form' will be filled.

All these evaluation stages will be done in the form of dividing 171 patients into 3 groups and evaluating them sequentially by numbering.

Application of manual hand massage: The researcher will receive certified training on hand massage. Hand massage application method will be determined after the training.

Application of machine-based hand massage: The pressure of the machine will be adjusted according to the manual massage application method. In manual massage and machine massage, machine adjustments will be made to keep the temperature and pressure difference as low as possible.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Having undergone laparoscopic cholecystectomy,
* No complications after laparoscopic cholecystectomy,
* Receiving analgesia treatment according to the clinical protocol,
* Pain score >4 according to the Numerical Rating Scale,
* Able to speak and understand Turkish
* No visual or auditory problems,
* No diagnosed psychiatric problem,
* No diagnosed gastrointestinal problem,
* Voluntary patients will be included.

Exclusion Criteria:

* Having undergone open cholecystectomy,
* Complications after laparoscopic cholecystectomy,
* Pain score ≤4 according to the Numerical Rating Scale,
* Using analgesic drugs or methods other than clinical protocol,
* Having visual or auditory problems,
* Having a diagnosed psychiatric problem,
* Diagnosed gastrointestinal problem,
* Patients with contagious skin disease (such as zoster, fungus, wart, eczema) on their hands, presence of thrombosis or phlebitis, any fracture, ligament injury,
* Non-voluntary patients will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) before the massage. A score of 0-10 is given on the NRS. A score of 0 on NRS means I have no pain. A score of 10 means I have unbearable pain.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) after the hand massage applied at the 0th hour. A score of 0-10 is given on the NRS. A score of 0 on NRS means no pain. 10 points means unbearable pain.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) after the hand massage applied at the 4th hour. A score of 0-10 is given on the NRS. A score of 0 on NRS means no pain. 10 points means unbearable pain.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) after the hand massage applied at the 8th hour. A score of 0-10 is given on the NRS. A score of 0 on NRS means no pain. 10 points means unbearable pain.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) before the massage. A score of 0-10 is given on the NRS. A score of 0 on NRS means I have no pain. A score of 10 means I have unbearable pain.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) after the hand massage applied at the 0th hour. A score of 0-10 is given on the NRS. A score of 0 on NRS means no pain. 10 points means unbearable pain.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) after the hand massage applied at the 4th hour. A score of 0-10 is given on the NRS. A score of 0 on NRS means no pain. 10 points means unbearable pain.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | It will be evaluated using the numerical rating scale (NRS) after the hand massage applied at the 8th hour. A score of 0-10 is given on the NRS. A score of 0 on NRS means no pain. 10 points means unbearable pain.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | Immediately after surgery, it will be evaluated using the numerical rating scale. A score of 0-10 is given on the NRS. A score of 0 on NRS means I have no pain. A score of 10 means I have unbearable pain.
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | After surgery at 0 hour it will be evaluated using a numerical rating scale. A score of 0-10 is given on the NRS. A score of 0 on NRS means I have no pain. A score of 10 means I have unbearable pain.
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | After surgery at 4 hour it will be evaluated using a numerical rating scale. A score of 0-10 is given on the NRS. A score of 0 on NRS means I have no pain. A score of 10 means I
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Pain After Laparoscopic Cholecystectomy Surgery | After surgery at 8 hour it will be evaluated using a numerical rating scale. A score of 0-10 is given on the NRS. A score of 0 on NRS means I have no pain. A score of 10 means I
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used immediately after the surgery and before the massage to be performed at the 0th hour.
  To see the effect of manual hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used after the massage performed at the 0th hour after the surgery.
  To see the effect of manual hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used after the massage performed at the 4th hour after the surgery.
  To see the effect of manual hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used after the massage performed at the 8th hour after the surgery.
  To see the effect of manual hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The Trait Anxiety Scale is used. The Trait Anxiety Scale will be used once before the surgery.
  To see the effect of manual hand massage on trait anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used immediately after the surgery and before the massage to be performed at the 0th hour.
  To see the effect of machine-based hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used after the massage performed at the 0th hour after the surgery.
  To see the effect of machine-based hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used after the massage performed at the 4th hour after the surgery.
  To see the effect of machine-based hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The State Anxiety Scale is used. The State Anxiety Scale will be used after the massage performed at the 8th hour after the surgery.
  To see the effect of machine-based hand massage on state anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The Trait Anxiety Scale is used. The Trait Anxiety Scale will be used once before the surgery.
  To see the effect of machine-based hand massage on trait anxiety level
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | Immediately after surgery the State Anxiety Scale is used.
  Evaluation of state anxiety level of patients who were not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | After surgery at 0th hour the State Anxiety Scale is used.
  Evaluation of state anxiety level of patients who were not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | After surgery at 4th hour the State Anxiety Scale is used.
  Evaluation of state anxiety level of patients who were not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | After surgery at 8th hour the State Anxiety Scale is used.
  Evaluation of state anxiety level of patients who were not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Anxiety After Laparoscopic Cholecystectomy Surgery | The Trait Anxiety Scale is used. The Trait Anxiety Scale will be used once before the surgery.
  Evaluation of trait anxiety level of patients who were not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. Before the massage, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. After the hand massage applied at 0th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. After the hand massage applied at 4th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. After the hand massage applied at 8th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of manual hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. Before the massage, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. After the hand massage applied at 0th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. After the hand massage applied at 4th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | The form of monitoring of gastrointestinal functions is used. After the hand massage applied at 8th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  To see the effect of machine-based hand massage
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | immediately after surgery, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | After surgery at 0th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | After surgery at 4th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  assessing patients who are not massaged (control group)
The Effect of Machine-Based and Manually Applied Hand Massage on Gastrointestinal System Functions After Laparoscopic Cholecystectomy Surgery | After surgery at 8th hour, it will be evaluated using a The form of monitoring of gastrointestinal functions.
  assessing patients who are not massaged (control group)

CONTACTS AND LOCATIONS:
Overall Officials: Münevver Şengül, Principal Investigator — mnvvrsngll58@gmail.com; Sevim Çelik, Study Director — sevimakcel@yahoo.com
Locations (1):
- Bartin universty, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No